CLINICAL TRIAL: NCT05738317
Title: A Prospective, Single-arm, Phase II Trial of Adebrelimab Combined With Bevacizumab and Albumin Paclitaxel in Advanced Non-squamous Non-small Cell Lung Cancer After First-line Immunotherapy Progression
Brief Title: Adebrelimab Combined With Bevacizumab and Albumin Paclitaxel in Non-squamous NSCLC After First-line Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiaorong Dong (Other)
Responsible Party: Sponsor-Investigator, Xiaorong Dong, Professor/Chief Physician, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-NSCLC-II-026
Record Dates: First submitted 2023-02-12; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab

STUDY DESIGN:
Intervention Model Description: Patients with advanced non-squamous non-small cell lung cancer after first-line immunotherapy progression
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adebrelimab Combined With Bevacizumab and Albumin Paclitaxel (Experimental): Adebrelimab: 20 mg/kg Adebrelimab is given on day 1 of each cycle, with 1 dosing cycle every 3 weeks. The dosing time window may be ±5 days, but within 72 hours before each dose, subjects must complete an examination including all clinically necessary tests to assess tolerability of continued dosing, in addition to imaging. Subjects are also advised to remain in the hospital for observation 72 hours after the first dose.
  Bevacizumab: 7.5 mg/kg Bevacizumab administered intravenously on day 1 of each cycle, with 1 dosing cycle every 3 weeks.
  Albumin Paclitaxel: 100 mg/m2 Albumin Paclitaxel is given on days 1, 8, and 15 of each cycle by intravenous infusion for 1 dosing cycle every 3 weeks.
  Interventions: Drug: Adebrelimab Combined With Bevacizumab and Albumin Paclitaxel

INTERVENTIONS:
Drug: Adebrelimab Combined With Bevacizumab and Albumin Paclitaxel — Adebrelimab is recommended to be administered with an infusion pump. The infusion pipeline is equipped with a 0.22-micron online filter membrane. Intravenous injection or bolus injection is not allowed. At the end of infusion, flush the infusion tube with sufficient 5% glucose or physiological saline, and do not share the same infusion tube with other drugs. In each treatment cycle, Adebrelimab should be given intravenously first.

SUMMARY:
A prospective, single-arm, phase II trial of Adebrelimab combined with bevacizumab and albumin paclitaxel in advanced non-squamous non-small cell lung cancer after first-line immunotherapy progression.

DETAILED DESCRIPTION:
The study consisted of a screening period (no more than 4 weeks after patients signed informed consent until enrollment, with imaging assessments allowed to be archived within 4 weeks prior to enrollment), a treatment period (treatment termination defined as discontinuation of treatment for any reason, or withdrawal from the study for any reason), a safety follow-up period, and a survival follow-up period.

Screening period:

Patients were required to undergo a screening evaluation to determine their eligibility for the study within 4 weeks prior to enrollment.

Patients eligible for the study receive adebrelimab, 20 mg/kg, Intravenous infusion, Q3W + bevacizumab, 7.5 mg/kg, Intravenous infusion, Q3W + albumin paclitaxel 100 mg/m2, D1, 8, 15, Intravenous infusion, Q3W. albumin paclitaxel treatment for 4 cycles, adebrelimab, bevacizumab use to PD, intolerable toxicity, patient withdrawal of informed consent, investigator decision to discontinue study treatment.

Treatment period:

Patients eligible for study enrollment were given medication sequentially on day 1 of each cycle, with a dosing window of ±5 days, and patients were required to complete various examinations including vital signs, height and weight, physical examination, laboratory tests, and physical status scores to assess tolerance for continued treatment. The specific examinations and requirements for each visit are shown in the study flow chart.

End of treatment:

End of treatment is defined as confirmation of disease progression or withdrawal from the study and requires an end-of-treatment visit ±5 days from the time of the decision to discontinue treatment and/or withdraw from the study.

Safety follow-up. Safety follow-up visits will be conducted within 30±7, 60±7 days, and 90±7 days after the last dose.

Survival follow-up. Survival follow-up will be conducted every 3 months after safety follow-up and telephone follow-up is acceptable.

ELIGIBILITY:
Inclusion Criteria:

1. voluntarily enrolled in this study and signed the Informed Consent Form (ICF).
2. age ≥ 18 years and both sexes
3. patients with metastatic or recurrent stage IV non-squamous NSCLC (AJCC 8th edition TNM stage) proven by histopathological or cytopathological diagnosis, mainly including adenocarcinoma, large cell lung cancer, adenocarcinoma with squamous differentiation or adenosquamous carcinoma with predominantly adenocarcinoma component may also be enrolled if eligible by study assessment.
4. objective imaging progression (RECIST v1.1 assessment) after subjects have received a first-line regimen containing immune checkpoint inhibitor therapy.
5. the best outcome of first-line immune checkpoint inhibitor-containing therapy is SD, PR, CR, and PFS of ≥ 3 months on first-line therapy.
6. imaging evaluation (CT or MRI) with at least one measurable target lesion (according to RECIST v1.1 criteria) within 4 weeks prior to enrollment.
7. an ECOG PS score of 0-1 within 4 weeks prior to enrollment.
8. an expected survival of ≥ 12 weeks.
9. function of vital organs in accordance with the following requirements. (1) blood routine: white blood cell count (WBC) ≥ 3.0×109/L; absolute neutrophil count (ANC) ≥ 1.5×109/L; platelets (PLT) ≥ 100×109/L; hemoglobin level (HGB) ≥ 9.0 g/dL (no corresponding supportive treatment such as blood transfusion and leukocyte boosting within 7 days).

(2) Liver function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times ULN in patients without liver metastases, ALT and AST ≤ 5 times ULN in patients with liver metastases; serum total bilirubin (TBIL) ≤ 1.5 times ULN (except total bilirubin < 3.0 mg/dL in Gilbert syndrome); albumin (ALB) ≥ 30 g/L, alkaline phosphatase (ALP) ≤ 2.5×ULN, and in patients with bone metastases, ALP ≤ 5×ULN.

(3) renal function: serum creatinine ≤ 1.5 times ULN or creatinine clearance (CrCl) ≥ 50 mL/min (using Cockcroft/Gault formula); urine protein (UPRO) < (++), or 24-hour urine protein amount < 1.0 g.

(4) Coagulation function: international normalized ratio (INR) ≤ 1.5 and activated partial thromboplastin time (APTT) ≤ 1.5 times ULN; if the patient is receiving anticoagulation therapy, as long as PT or APTT is within the therapeutic range of the intended use of anticoagulants, referring to the relevant drug instructions.

(5) Thyrotropin (TSH) ≤ upper limit of normal (ULN); if abnormal, T3 and T4 levels should be examined; normal T3 and T4 levels are eligible for enrollment.

10. Non-surgical sterilization or female patients of childbearing age must have a negative serum pregnancy test within 7 days prior to the first dose and must be non-lactating. Female patients of childbearing age or male patients whose partners are women of childbearing age must agree to use highly effective methods of contraception during the study period and for 6 months after the last administration of the study drug.

Exclusion Criteria:

1. patients with other pathological tissue types of non-small cell lung cancer (including squamous cell carcinoma, mixed non-small cell and small cell lung cancer, and predominantly squamous adenosquamous carcinoma of the lung)
2. patients with known EGFR-sensitive mutations (19Exon del/21Exon L858R), positive ALK/ROS1 fusion, BRAFV600E mutation, MET gene exon 14 jump mutation, positive RET gene fusion, and other patients with approved targets for targeted agents.
3. patients with imaging showing signs of tumor invasion into the great vessels, where the tumor has completely approached, encircled, or invaded the lumen of a great vessel (e.g., pulmonary artery or superior vena cava)
4. patients with hypertension whose blood pressure is not satisfactorily controlled by antihypertensive medication (sitting systolic blood pressure > 150 mmHg, or diastolic blood pressure > 100 mmHg), previous hypertensive crisis or hypertensive encephalopathy
5. those with a known hereditary bleeding tendency or coagulation disorders; those who have received full-dose anticoagulant or thrombolytic therapy within 10 days prior to enrollment, or those who have taken non-steroidal anti-inflammatory drugs with platelet inhibitory effects within 10 days prior to enrollment (except for prophylactic use of low-dose aspirin (≤325 mg/day)).
6. had a hemoptysis of 2nd degree or greater with a single hemoptysis of ≥1/2 teaspoon (2.5 ml) within 3 months prior to enrollment
7. thrombosis in the 6 months prior to enrollment and an arterial/venous thrombotic event within 1 year prior to screening, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis, and pulmonary embolism.
8. those with severe vascular lesions (including aneurysms or arterial thrombosis requiring surgical treatment) within 6 months prior to enrollment
9. late first-line treatment with anti-angiogenic agents, including but not limited to bevacizumab, apatinib, anlotinib, ramucirumab, lenvatinib, etc.; treatment with paclitaxel, including paclitaxel, albumin paclitaxel, paclitaxel liposome, docetaxel (polyene paclitaxel), etc;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
6-month PFS rate | 6 months
  6-Month PFS Rates for Adebrelimab Combined with Bevacizumab and Albumin Paclitaxel in Patients with Advanced NSCLC Progressed by First-Line Immunotherapy Evaluated by Investigators

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 12 months
  PFS is defined as the time elapsed between the start of treatment and the first sign of disease progression or death from any cause.
Over survival (OS) | up to 12 months
  OS is defined as the time elapsed between the initiation of treatment and mortality from any cause.
Disease control rate (DCR) | up to 12 months
  Number of cases with completed/partial response and stable disease after treatment as a percentage of evaluable cases.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaorong Dong, Dr., Study Chair — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.